CLINICAL TRIAL: NCT02169375
Title: Effect of Normalizer Adaptation on Accuracy in a Sensorimotor Based Brain-Computer Interface
Brief Title: Sensorimotor Based Brain Computer Interface
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient improvement in primary measures under either condition.
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jane Huggins, PhD, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: I0004; R21HD054913 (NIH)
Record Dates: First submitted 2014-06-16; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mu Rhythm with adaptation (Experimental)
  Interventions: Other: Brain computer Interface Mu (SMR) rhythm
- Mu Rhythm without adaptation (Experimental)
  Interventions: Other: Brain computer Interface Mu (SMR) rhythm

INTERVENTIONS:
Other: Brain computer Interface Mu (SMR) rhythm — Subjects will wear an EEG cap for 1-2 hours typical per session and use the brain computer interface to operate assistive technology. Subjects will be asked to participate in 10 sessions.

SUMMARY:
Sensorimotor (also know as mu) rhythm based brain-computer interfaces (BCIs) are a tool for controlling electronic devices using only brain signals. Often, the computer software that analyzes mu-rhythm brain signals constantly adapts to the individual user's brain signals when the training target location is known. The investigators want the BCIs to be more universal, and not depend on knowing the target location. Therefore, the investigators will test the effect removing adaptation has on accuracy of using a mu-rhythm BCI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Able to read text on a computer screen
* Able to understand and remember instructions concerning participation.

Exclusion Criteria:

* Unable give informed consent.
* Unable to understand and follow instructions.
* Have abnormal tone or uncontrolled movements in the head-and-neck that would interfere with EEG recordings.
* Known to have photosensitive epilepsy.
* Open head lesions or sores.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Accuracy of a mu rhythm BCI using adaptation versus no adaptation. | 10 times over 5 weeks
  Accuracy with which subjects can select one of two targets after a 3-second time period. The accuracy for a run is calculated as the % of the trials in which the correct target is selected. The average accuracy will be calculated for each of the 10 usage sessions and changes over the sessions will be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Huggins, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States